CLINICAL TRIAL: NCT00833599
Title: Phase I/II Combinational Investigational New Drug Application: Imaging Lymphatic Function in Normal Subjects and in Persons With Lymphatic Disorders
Brief Title: Imaging Lymphatic Function in Normal Subjects and in Persons With Lymphatic Disorders
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Cancer Institute (NCI) (NIH); Lymphatic Malformation Institute (Other); Lipedema Foundation (Other)
Responsible Party: Principal Investigator, Eva Sevick, Professor of Molecular Medicine; Director of Center for Molecular Imaging, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-IMM-08-0415; R01HL092923 (NIH); R01CA128919 (NIH)
Record Dates: First submitted 2009-01-30; First posted 2009-02-02 (Estimated); Last update posted 2018-05-23 (Actual); Status verified 2018-05

CONDITIONS: Lymphedema; Lymphatic Disorders; Lipedema; Vascular Malformation; Vascular Anomaly; Dercum Disease
Keywords: Lymphedema; Genetic; Lymphatic Disorder; Lipedema; Vascular Malformation; Vascular Anomaly; Dercum Disease
MeSH Terms: conditions — Lymphedema; Lymphatic Diseases; Lipedema; Vascular Malformations; Adiposis Dolorosa | interventions — Indocyanine Green

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — DNA from blood or saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: NIRFLI with ICG: 1) Persons affected with lymphatic or lympho-vascular disorders, 2) Family members (affected or unaffected) of persons affected with lymphatic or lympho-vascular disorders and 3) Health, normal persons (Controls) that participate at one of the clinical sites in both the lymphatic function imaging with indocyanine green and the Near-infrared Fluorescence Lymphatic Imaging (NIRFLI) system, as well, as the genetic analysis portion of the study.
  Interventions: Drug: NIRFLI with ICG
- 2: Genetic Analysis Only: Family members of an affected subject from Group 1. Subjects in Group 2 can be either affected or unaffected and will provide a blood or saliva sample for the genetic analysis portion of the study, but will not undergo lymphatic function imaging with ICG and the NIRFLI system. Group 2 individuals are not required to travel to one of the clinical sites in order to participate in the study.

INTERVENTIONS:
Drug: NIRFLI with ICG — We conduct Near-infrared Fluorescence Lymphatic Imaging following the off-label use of Indocyanine Green as a lymph contrast agent and the use of a custom designed fluorescence imager to dynamically follow lymphatic trafficking in subjects. We seek to use the resulting phenotypes acquired in normal and diseased patients to correlate to mutations of specific genes reported to be associated with lymphatic development.
  Other Names: IC-Green; Cardio-Green; ICG; Near-infrared Fluorescence Lymphatic Imaging (NIRFLI)
  Groups: 1: NIRFLI with ICG

SUMMARY:
The purpose of this study is to demonstrate the feasibility of near-infrared fluorescence imaging in subjects with acquired or hereditary lymphedema, in subjects with lipidema and other lymphovascular disorders and in normal health subjects; in order to attempt to correlate imaging phenotype(s) with genotype(s).

DETAILED DESCRIPTION:
Currently, there is no method to assess lymphatic function in persons with acquired (developed following surgery or trauma) lymphedema, hereditary lymphedema or other lympho-vascular disorders. The causes of these disorders, and the means to distinguish between them, is not available from existing diagnostics. A method to monitor lymphatic function could assist in the development of new therapies, the prediction of a patient's susceptibility to develop these disorders, and the evaluation of patient's conditions or responses to therapy and treatment. In this Phase I/II trial, we inject Indocyanine Green (ICG) off-label as a lymph contrast agent and use a custom designed fluorescence imager to conduct near-infrared fluorescence imaging to dynamically follow lymphatic trafficking in subjects. Blood is also collected for DNA analysis. The resulting images are analyzed, and the phenotypes observed in both normal and diseased subjects are used to correlate to mutations of specific genes reported to be associated with lymphatic development.

ELIGIBILITY:
Inclusion Criteria for Participation in NIRFLI with ICG (Group 1):

1. Negative urine pregnancy test within 36 hours prior to study drug administration, if female of childbearing potential.
2. Females must complete the Female Enrollment Form. Those subjects of childbearing potential must agree to use one of the medically accepted methods of contraception listed on the form for a period of one month following the study. Female subjects of non-childbearing potential, defined as physiologically incapable of becoming pregnant, must meet the criteria listed on the Female Enrollment form, but are not restricted to the use of contraception following study participation.
3. Subjects must be able to lie on their backs for periods of 10 minutes at at time for up to a total of 60 minutes.
4. Children must be able to remain reasonably still for the time required for imaging.
5. Subjects with lymphatic dysfunction must be diagnosed with lymphedema, lipedema, or vascular malformation/anomaly that suggests a lymphatic component.

Exclusion Criteria for Participation in NIRFLI with ICG (Group 1):

1. Persons with mobililty issues that could make participating too difficult
2. Women who are pregnant or breast-feeding
3. Persons who are allergic to iodine
4. Persons who weigh in excess of 400 lbs
5. If the subject is a female of child-bearing potential, she must agree to use a contraceptive for one month after study participation.
6. Persons who do not meet inclusion criteria.

Inclusion Criteria for Participation in Genetic Analysis Only (Group 2):

1. The subject has a family member with lymphatic dysfunction.
2. The subject is willing to have blood drawn or saliva collected for DNA analysis

Exclusion Criteria for Participation in Genetic Analysis Only (Group 2):

1) The subject has experienced a medical problem from a prior blood draw

Min Age: 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 1) Persons with lymphatic dysfunction (e.g. lymphedema, lipedema, dercums, etc.), 2) Persons with vascular malformation that suggest a lymphatic component, 3) Family members of persons, whom participated in this study, with a lymphatic dysfunction or vascular malformation that suggests a lymphatic component and 3) Healthy, normal individuals as controls
Sampling Method: Non-Probability Sample
Enrollment: 283 (Estimated)
Dates: Start 2009-01; Primary Completion 2019-12 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Near-infrared fluorescence lymphatic imaging (NIRFLI) provides informaton on lymphatic function or dysfunction to diagnose disorders | Images are collected for up to 3 hours after injection with indocyanine green

CONTACTS AND LOCATIONS:
Overall Officials: Eva M Sevick, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (3):
- United States (3):
  - Lymphedema Clinic at Memorial Hermann Hospital in the Texas Medical Center, Houston, Texas
  - UT Physicians Pediatric Surgery Clinic, Houston, Texas
  - Wound Care Clinic at CHI St. Luke's The Woodland's Hospital, The Woodlands, Texas

REFERENCES:
- [Background] Rasmussen JC, Tan IC, Marshall MV, Fife CE, Sevick-Muraca EM. Lymphatic imaging in humans with near-infrared fluorescence. Curr Opin Biotechnol. 2009 Feb;20(1):74-82. doi: 10.1016/j.copbio.2009.01.009. Epub 2009 Feb 23. PMID 19233639
- [Derived] Rasmussen JC, Zvavanjanja RC, Aldrich MB, Greives MR, Sevick-Muraca EM. Near-infrared fluorescence lymphatic imaging of Klippel-Trenaunay syndrome. J Vasc Surg Venous Lymphat Disord. 2017 Jul;5(4):533-537. doi: 10.1016/j.jvsv.2017.01.011. PMID 28623992